CLINICAL TRIAL: NCT04123808
Title: Dosing Effects of an Upper Extremity Rehabilitation Program Using a Brain-Computer Interface Mediated Robotic Hand Orthosis for Chronic Stroke Patients: IpsiHand System
Brief Title: IpsiHand System for Rehabilitation of the Arm and Hand After Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by sponsor
Sponsor: Columbia University (Other)
Collaborators: Neurolutions, Inc. (Industry)
Responsible Party: Principal Investigator, Joel Stein, MD, Professor and Chair of the Department of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS4076
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Hemiparesis; Rehabilitation; Upper Extremity; Neurological Rehabilitation; Neuronal Plasticity; Brain-Computer Interfaces; Robotics
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Masking Description: An occupational therapist independent to the study will review and score 2 outcome measures (Fugl-Meyer and Action Research Arm Test). The study coordinator will randomize the order of the videos for each participant, so that the outcome assessor will not know which time point they are scoring. In other words, the video-outcome assessor will be blinded to the order of the assessments as they are scoring them but will not be blinded to the intervention as all participants will be receiving the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- IpsiHand Treatment (Experimental): All participants will receive treatment with IpsiHand device
  Interventions: Device: IpsiHand Treatment

INTERVENTIONS:
Device: IpsiHand Treatment — The IpsiHand system utilizes a Brain-Computer Interface (BCI) as a control for a robotic hand orthosis donned on the affected upper extremity as participants are guided through a rehabilitation program on a tablet. Participants will complete 16-32 weeks of home therapy with the IpsiHand system. Motor function of their impaired upper extremity will be evaluated at baseline, at 4-week intervals, and 3 months post no-device use, to track progress.

SUMMARY:
This study aims to assess whether the NeuroLutions Upper Extremity Rehabilitation System (known as IpsiHand) will help stroke patients regain strength and functional movements in their arm. The IpsiHand system involves using a hand robotic device that is controlled by brain waves, known as a Brain-Computer Interface (BCI). By using the device, participants will be harnessing brainwaves from the side of their brain not affected by stroke to control the robotic device on the hand that is weaker from the stroke.

DETAILED DESCRIPTION:
This trial aims to assess the effectiveness of the NeuroLutions Upper Extremity Rehabilitation System, known as IpsiHand, on functional motor recovery and neuroplasticity for chronic stroke survivors with hemiparesis (N=27). The IpsiHand system involves a Brain-Computer Interface (BCI) as a control for a robotic hand orthosis. Participants will complete 16-32 weeks of home therapy with the IpsiHand system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke(s), with most recent stroke at least 6 months prior to study start (can be ischemic or hemorrhagic)
* PROM: Full extension of digits 2 and 3 at MPs, PIPs, and DIPs
* English speaking
* Intact cognition to provide informed consent
* Intact language skills to comprehend and follow directions
* Experiencing difficulty performing ADLs with affected upper limb
* Upper extremity Botox allowable, but not required

  * Botox users must continue regimen at regular intervals for duration of study
  * Botox users will provide clinic note for each injection (date, dose, and muscle location)
  * Botox + Study Schedule
* At study initiation, Botox injection will occur between 3-7 days prior to baseline measurement and initiation of device use
* Repeat Botox injections must be completed at least 3 days prior to any administration of the outcome measures

Exclusion Criteria:

* Concurrent participation in another study
* Co-morbid orthopedic condition/pain limiting functional use of the impaired upper limb
* History of neurological disorder other than stroke
* Botox user unable to comply with above noted requirements
* Ongoing physical or occupational therapy addressing the upper limb
* Ongoing electric stimulation or other rehabilitative devices (e.g. robotics, virtual reality) to upper limb
* Cognitive impairment: Short Blessed Test Score 9
* Significant spasticity: Modified Ashworth Scale score 3 at the elbow
* Significant hemispatial neglect: Mesulam Cancellation Test 3 unilaterally
* Insufficient Strength: Motricity Index score for shoulder abduction 18
* Significantly impaired sensation of impaired upper limb: National Institutes of Health Stroke Scale - Item 8 (Sensory) score of 2
* History of cranioplasty
* History of seizure disorder
* No changes to usual exercises, splint use, or oral baclofen/anti-spasticity medication use during trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Motor Recovery after Stroke for Upper Extremity | Baseline through 3 months post no device use
  The Fugl-Meyer is a scale that measures capacity of the arm. There are 33 items that evaluate reflexes, active movement, grasp patterns, speed, and coordination of the arm and hand. Each item is scored from 0-2, with a maximum total score of 66. Higher scores indicate better performance.

SECONDARY OUTCOMES:
Action Research Arm Test | Baseline through 3 months post no device use
  The ARAT is a scale that measures activity participation of the arm. There are 19 items that several types of grasps, grips, pinches, and gross movements of the arm and hand. Each item is scored from 0-3, with a maximum total score of 57. Higher scores indicate better performance.
Box and Block Test | Baseline through 3 months post no device use
  The Box and Block Test measures the number of blocks a participant can pick up and place over a patrician in 1 minute. The number of blocks successfully moved are counted and a higher number indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bundy DT, Souders L, Baranyai K, Leonard L, Schalk G, Coker R, Moran DW, Huskey T, Leuthardt EC. Contralesional Brain-Computer Interface Control of a Powered Exoskeleton for Motor Recovery in Chronic Stroke Survivors. Stroke. 2017 Jul;48(7):1908-1915. doi: 10.1161/STROKEAHA.116.016304. Epub 2017 May 26. PMID 28550098
- [Background] Cervera MA, Soekadar SR, Ushiba J, Millan JDR, Liu M, Birbaumer N, Garipelli G. Brain-computer interfaces for post-stroke motor rehabilitation: a meta-analysis. Ann Clin Transl Neurol. 2018 Mar 25;5(5):651-663. doi: 10.1002/acn3.544. eCollection 2018 May. PMID 29761128
- [Background] Zeiler SR, Krakauer JW. The interaction between training and plasticity in the poststroke brain. Curr Opin Neurol. 2013 Dec;26(6):609-16. doi: 10.1097/WCO.0000000000000025. PMID 24136129